CLINICAL TRIAL: NCT06565650
Title: A Randomized, Multicenter, Double-Masked, Saline-Controlled Trial to Evaluate Corneal Endothelial Cell Density in Subjects With Dry Eye Disease Administering Miebo® (Perfluorohexyloctane Ophthalmic Solution) for 12 Months.
Brief Title: A Study to Evaluate Corneal Endothelial Cell Density (ECD) in Subjects With Dry Eye Disease (DED) Administering Miebo® (Perfluorohexyloctane Ophthalmic Solution) for 12 Months.
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 933
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — perfluorohexyl-octan; Sodium Chloride

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Subjects will be instructed not to show or discuss the properties of the assigned Investigational Product (IP) and/or their experience with the IP with other subjects and not to show or discuss the IP with the Investigator or site personnel other than the dedicated dosing coordinator, unless instructed to do so.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Miebo (Experimental): 100% perfluorohexyloctane 4 times daily (QID)
  Interventions: Drug: Miebo
- Saline solution (Placebo Comparator): (0.6% sodium chloride solution) 4 times daily (QID)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Miebo — 100% perfluorohexyloctane
  Arms: Miebo
Drug: Saline — 0.6% sodium chloride solution
  Arms: Saline solution

SUMMARY:
A Randomized, Multicenter, Double-Masked, Saline-Controlled Trial to Evaluate Corneal Endothelial Cell Density in Subjects With Dry Eye Disease Administering Miebo® (Perfluorohexyloctane Ophthalmic Solution) for 12 Months

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 18 years of age at the time of consent.
2. Have a self-reported history of DED in both eyes (OU) for at least 6 months prior to Visit 1 (Screening/Baseline)
3. Have a total corneal fluorescein staining score (tCFS) score >2 in both eyes
4. Have an Ocular Surface Disease Index (OSDI) score >17
5. Have a baseline ECD ≥1750 cells/mm2 in each eye
6. Provide written informed consent
7. Be able and willing to follow instructions, including participation in all trial assessments and visits
8. If a contact lens wearer, be willing to discontinue contact lens use during and for 30 minutes following instillation of investigational drug and during study visits

Exclusion Criteria:

1. Be at least 18 years of age at the time of consent.
2. Have a self-reported history of DED in both eyes (OU) for at least 6 months prior to Visit 1 (Screening/Baseline)
3. Have a total corneal fluorescein staining score (tCFS) score >2 in both eyes
4. Have an Ocular Surface Disease Index (OSDI) score >17
5. Have a baseline ECD ≥1750 cells/mm2 in each eye
6. Provide written informed consent
7. Be able and willing to follow instructions, including participation in all trial assessments and visits
8. If a contact lens wearer, be willing to discontinue contact lens use during and for 30 minutes following instillation of investigational drug and during study visits
9. Have any clinically significant ocular surface slit lamp findings and/or in the opinion of the Investigator have any findings that may interfere with trial parameters in either eye
10. Have an ocular or periocular malignancy in either eye
11. Have a history of herpetic keratitis in either eye
12. Have any planned ocular and/or lid surgeries in either eye during the course of the study
13. Have a known allergy and/or sensitivity to the IP
14. Have a history of ocular laser surgery in either eye within 3 months (90 days) prior to Visit 1 (Screening/Baseline)
15. Have a history of incisional ocular surgery or severe trauma in either eye within 3 months (90 days) prior to Visit 1 (Screening/Baseline)
16. Have high contrast best-corrected visual acuity equal to or worse than logMAR +0.7 (Snellen equivalent score of 20/100 or worse) as assessed by Early Treatment Diabetic Retinopathy Study (ETDRS) scale in either eye, obtained under bright room lighting
17. Be a woman who is pregnant, nursing or planning a pregnancy during the course of the study
18. Be a woman of childbearing potential who is unwilling to submit to a urine pregnancy test. Non-childbearing potential is defined as a woman who is permanently sterilized (eg, has had a hysterectomy or bilateral tubal ligation or bilateral oophorectomy) or is postmenopausal (without menses for 12 consecutive months).
19. Be a woman of childbearing potential who is not using an acceptable method of birth control. Acceptable methods of contraception include hormonal - oral, implantable, injectable, or transdermal - contraceptives; mechanical contraception - spermicide in conjunction with a barrier such as a diaphragm or condom; intrauterine device; or surgical sterilization of partner. For non-sexually active females, abstinence may be regarded as an adequate method of birth control; however, the subject must agree to use adequate birth control as defined above for the remainder of the study if she becomes sexually active during the trial.
20. Be currently enrolled in an investigational drug or device trial or plan to enroll during the course of the study
21. Have a condition or be in a situation that the Investigator believes may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2024-07-31 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in ECD | Assessed at Month 3 and Month 12 Visits
  Mean change from baseline in ECD in the study eye at the Month 3 and Month 12 Visits

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Site 101, Glendale, California
  - Site 112, Murrieta, California
  - Site 102, Newport Beach, California
  - Site 109, Rancho Cordova, California
  - Site 106, Torrance, California
  - Site 113, Delray Beach, Florida
  - Site 107, Morrow, Georgia
  - Site 105, Carmel, Indiana
  - Site 110, Kansas City, Missouri
  - Site 104, St Louis, Missouri
  - Site 108, Asheville, North Carolina
  - Site 103, Memphis, Tennessee